CLINICAL TRIAL: NCT06320314
Title: Evaluation of the Efficacy and Tolerability of the Tested Formula 2039125 03 BID After 3 Months in the Treatment of Facial Hyperpigmentation of 3 Origins: Melasma, Acne Induced Post-Inflammatory Hyperpigmentation and Solar Lentigo
Brief Title: Efficacy and Tolerability of Tested Formula After 3 Months in Treatment of Facial Hyperpigmentation of 3 Origins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LRP23021-E serum
Record Dates: First submitted 2024-03-11; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hyperpigmentation
Keywords: facial hyperpigmentation; melasma; acne induced PIHP; solar lentigo
MeSH Terms: conditions — Hyperpigmentation; Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mild to moderate melasma (Experimental): adult patients suffering from mild to moderate melasma (Investigator's Global Assessment (IGA) 1 or 2)
  Interventions: Other: tested product (2039125 03)
- mild to moderate acne induced PIHP (Experimental): adult patients suffering from mild to moderate acne-induced PIHP (IGA 1 or 2) without active acne (i.e., less than 10 inflammatory lesions)
  Interventions: Other: tested product (2039125 03)
- solar lentigo (Experimental): adult patients suffering from solar lentigo with a pigmentation score > 5
  Interventions: Other: tested product (2039125 03)

INTERVENTIONS:
Other: tested product (2039125 03) — application twice a day of the tested product (in the morning and evening) and a sunscreen (in the morning and at midday) to the face for 3 months

SUMMARY:
The objective of this study is to evaluate the efficacy, cosmetic acceptability and improvement of the stigmatization of the tested product (2039125 03) used bis in die (BID) for 3 months in adult patients suffering from mild to moderate melasma, or mild to moderate acne induced post-inflammatory hyperpigmentation, or solar lentigo.

DETAILED DESCRIPTION:
Hyperpigmentation is a common skin condition in which the colour of the skin becomes darker. These changes result from an excess of melanin production, distribution, or transport which can be caused by various internal and external factors such as genetic predisposition, hormonal changes, inflammation, acne, ultraviolet (UV) exposure.

Typical hyperpigmentation disorders include post-inflammatory hyperpigmentation, melasma and solar lentigines.

This open, single-centre, three-arm study is carried out with a new cosmetic formulation developed with the aim of acting on facial hyperpigmentation and used under normal conditions of use with before/after comparisons.

This clinical trial is conducted in accordance with the protocol, the HELSINKI declaration (1964) and subsequent amendments, and/or the International Council on Harmonization (ICH) Good Clinical Practices (GCP)/ and in compliance with applicable regulatory requirements.

Statistical Analysis:

* Efficacy Analysis: in each group, the quantitative parameters are analyzed using a mixed-effect model. This model includes Time and baseline as fixed effects. Patient are added as random effect. The comparisons between post-baseline time-point and baseline are performed whatever the interaction results using a Dunnett adjustment. Degrees of freedom for the comparisons are approximated by the Kenward-Roger method.
* Safety Analysis: no statistical analysis will be performed on safety. The data are presented descriptively.

Categorical data are summarized using the number and percentage of patients in each category. Continuous data are summarized using the arithmetic mean, Standard Deviation (SD), Q1, Q3, minimum, median and maximum values.

Regarding the sample size determination, there was no formal calculation. A number of 20 patients in each group (i.e. 60 patients in total) was considered sufficient to meet the study objective.

ELIGIBILITY:
Inclusion Criteria:

* all phototypes
* only one of the following pigmentary conditions on the face: epidermal or mixed, mild to moderate melasma; mild to moderate acne-induced PIHP; solar lentigo
* female patient of childbearing potential must use one of the reliable methods of contraception and agree not to change it during the study.

Exclusion Criteria:

* female patient who gave birth less than 3 months prior to Day 0, who is pregnant, breast-feeding or who plans to become pregnant during the study
* male patient with beard or facial hair, which would interfere with clinical evaluation or clinical procedure baseline)
* patient with any inflammatory dermatosis of the face such as seborrheic dermatitis, rosacea etc.
* severe melasma, dermal melasma
* patient with facial pigmentary disorders other than those described in inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
IGA score for patients with melasma or acne induced post-inflammatory hyperpigmentation (PIHP) | from baseline to Day84
  the hyperpigmentation is measured on a scale from 0 (cleared, almost cleared) to 3 (markedly darker than the surrounding normal skin)
modified Melasma Area and Severity Index (mMASI) for patients with melasma | from baseline to Day 84
  the mMASI is calculated using 3 components: four regions of the face (forehead, right malar, left malar and chin); area of involvement for each region (using a scale from 0 to 6): darkness compared to the surrounding normal skin for each area (evaluated using a scale from 0 to 6)
Post-Acne Hyperpigmentation Index (PAHPI) | from baseline to Day 84
  The PAHPI score is the sum of all 3 weighted scores: median lesion size (from 2 [< 3mm] to 8 [> 10mm], median lesion intensity (from 3 [slightly darker than surrounding skin] to 9 [significantly darker than surrounding skin] and number of lesions (from 1 [1-15] to 5 [> 60]. Total score ranges from 6 to 22.

SECONDARY OUTCOMES:
colorimetry measurements | from baseline to Day84
  skin color is measured using the L*a*b* color space (L* represents lightness, a* its position between green and red, b* its position between blue and yellow).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Pinto, Principal Investigator — PhDTrials center
Locations (1):
- PhDTrials Center, Lisbon, Portugal